CLINICAL TRIAL: NCT04259489
Title: Effectiveness of Share Care Diabetes Management in Patients With Type 2 Diabetes
Brief Title: Effectiveness of SCDM in Patients With Type 2 Diabetes
Acronym: ESCDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Professor and Director, Department of Endocrinology, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-T2DM
Record Dates: First submitted 2020-01-14; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Diabetes Education and Management; Share Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomization, parallel, controlled study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional therapy group (No Intervention): All patients in the control group will receive routine diabetes management, including lifestyle education, health guidance, blood glucose monitoring and medicine adjustment and other treatments which conducted by the endocrinology medical team. After the inclusion visit, the patients will be randomized to Shared Care group or traditional therapy group. Compared to conventional diabetes education in the traditional therapy group, the Shared Care group provides patients with online services and continuous diabetes management and education through a mobile application. It also addresses that it is important for patients to meet regularly with diabetes multidisciplinary team for better results. The total observation period is 3 years for each patient. The visits will be done every 3 months.
- Shared Care group (Active Comparator): The Patients download the Shared Care mobile application and connect with the smart-glucometer BG1 to upload blood glucose dairy in real time. With patient's informed consent, his or her data from each visit will be collected and recorded for analysis. After the patient returns home from the clinic, they can communicate through the APP with online diabetes educators. According to protocol, online diabetes educators answer patients' questions, give suggestions on patients' diet and summarize patients' issues to physicians, who provide high level supervision.
  Interventions: Behavioral: Shared Care diabetes management

INTERVENTIONS:
Behavioral: Shared Care diabetes management — After the inclusion visit, the patients will be randomized to Shared Care group or traditional therapy group. Compared to conventional diabetes education in the traditional therapy group, the Shared Care group provides patients with online services and continuous diabetes management and education through a mobile application. It also addresses that it is important for patients to meet regularly with diabetes multidisciplinary team for better results. The total observation period is 3 years for each patient. The visits will be done every 3 months.
  Arms: Shared Care group

SUMMARY:
This is a prospective, randomization, parallel, controlled study, which conducted to evaluate the effectiveness and related influencing factors of the Shared Care multidisciplinary diabetes care model. Patients with T2DM involved in the Shared Care model pay regularly quarterly visit to a multidisciplinary team led by physician at outpatient clinic, and receive remote and systematic management and education online after going home. After at least one year follow-up, evaluate the glycemic achieving rate (HbA1c<7%), the diabetes self-management behavior change and the effect of online diabetes self-management support for patients of the Shared Care multidisciplinary diabetes care model.

DETAILED DESCRIPTION:
Diabetes is a complex, chronic illness requiring continuous medical care with multifactorial risk-reduction strategies beyond glycemic control. At present, about 114 million diabetics and 11.6% incidence rate of diabetes in China have produced huge chronic disease management pressure and created great challenges for China's limited medical resources. (1-5). Meanwhile, with population aging and increasing prevalence of obesity in China, the number of patients with diabetes mellitus, diabetes-related complications and related mortality are expected to further increase, which also indicates greater healthcare expenditure and socioeconomic burden. A multi-center, cross-sectional survey of outpatients conducted in 606 hospitals across China showed that the majority of patients with type 2 diabetes did not achieve the goal of HbA1c <7.0% (6). There are varieties of problems including inadequate patient education, inability to track the out-of-hospital situation of diabetes, and lack of effective patient follow-up and education between each visits (1-5). Many researches have proved that comprehensive diabetes management education can significantly improve the quality of life of patients, decrease the incidence and mortality of diabetes complications, and relieve the government's medical economic burden (7). Besides, A number of studies have shown that the early detection and comprehensive management of diabetes can prevent the occurrence of a variety of complications and decrease the disability rate and premature death rate of diabetes. Therefore, how to improve the current situation of diabetes control in China is very important and a real problem in front of every doctor, patient and health institution. According to the diabetes management guidelines published by American Diabetes Association(ADA) and the National Institutes of Health(NIH), continuous follow-up of patients, diabetes self-management education and support (DSME/S) combined with multidisciplinary team comprehensive management can be abled to achieve better management results, and it is also a more comprehensive and cost-effective way to manage diabetic patients (8-12). In order to support health professionals to improve medical efficiency and promote patients develop healthy lifestyle, Shared Care diabetes management model established and believe that it will provide a sustained and effective solution for improving the effectiveness of comprehensive management for patients and reducing the burden of national chronic disease management.

The Shared Care aims to provide patients with a continuous management model of omni-directional and lifelong care management, and to strengthen diabetes self-management education and supports (DSME/S), achieve better health outcomes and delay incidence and mortality of diabetic complications. The model consisted of a medical team that includes dietitians, diabetes educators, nurses and physical therapist led by physician, and provides comprehensive disease and health management for patients with diabetes through outpatient consultation and out-of-hospital online continuous management. The management strategy is adjusted and individualized based on patients' habit and situation. Compared with traditional diabetes outpatient settings, patients of Shared Care return to the hospital for regular follow-up every three months since the initial visit after the informed consent. For each follow-up, a comprehensive management plan is made by a multidisciplinary team, including doctor consultation, diabetes management, foot evaluation, fundus assessment, insulin injection assessment, exercise evaluation and guidance, etc. The patients download the Shared Care mobile application during the outpatient service and connect with the smart-glucometer BG1 to upload blood glucose dairy, blood pressure diary and food log in real time.

With patient's informed consent, Patient-related vital signs (such as height, weight, body mass index, blood pressure, waist, hips), laboratory indicators (including glycated hemoglobin, low-density lipoprotein, total cholesterol, triglycerides, kidney indicators such as urine microalbumin and creatinine Ratio, glomerular filtration rate), blood glucose records, online learning frequency and other data will be uniformly recorded and comprehensively analyzed.

All out-of-hospital online diabetes educators are qualified as registered nurses. Before the start of the study, the nurses should uniformly receive training and examination related to diabetes education in the Department of Endocrinology of Chaoyang Hospital. The main contents of online education include personalized assessment and suggestions on diet, hyperglycemia and hypoglycemia events, drug use and insulin preservation as directed by doctors, and on blood glucose monitoring and reminders for revisit every three months, etc. In case of special circumstances or prescription adjustment, online diabetes educators should follow the training process to summarize the patient's condition with the doctor on the same day or during the weekly regular outpatient clinic, or arrange additional subsequent visit of the patient, all online consultation process is carried out under the supervision of the doctor (the diabetes educator spends about 5 minutes a week to discuss the condition of special patients with the doctor according to the actual situation). The model enables both patients and medical teams to carry out real-time data sharing, intelligent analysis and remote monitoring, thus significantly improving management efficiency and releasing medical resources.

A series of preliminary studies had been conducted in Chaoyang Hospital since January 2018. mean age of patients enrolled was 54.69 ± 11.14 years; the duration of diabetes was more than 7.8 ±7.0 years, and more than 70% were complicated with hypertension and / or dyslipidemia. The baseline glycemic achieving rate of patients with a duration more than 10 years was less than 35%. After participated in the Shared Care management model, glycemic achieving rate of patients with diabetic was more than 75%. Compared with the baseline HbA1c 7.4±1.5%, patients HbA1c in the latest follow-up was 6.6 ±1.0%, with the average decreased of 0.8 ±1.6% (P <0.05). The 3B achieving rate (HbA1c <7%, LDL-C < 2.6mmol/L, BP <130/80mmHg) of patients under the management of Shared Care Model was 21.84%. The baseline urinary microalbuminuria / creatinine (UACR) 35.8mg/g was not significantly increased compared with the last follow-up of 32.1mg/g (P>0.10). The daily cost of hypoglycemic medicine was significantly reduced in patients with the duration of diabetes less than 2 years or 15 years or more (medicine daily cost of the baseline and the latest follow-up was 3.5 RMB per day and 2.3 RMB per day respectively in patients with the duration of diabetes less than 2 years (P<0.05); medicine daily cost of the baseline and the latest follow-up was 10.4 RMB per day and 9.5 RMB per day respectively in patients with the duration of diabetes of 15 years or more (P<0.05)), but there was no significant increase in patients with other durations of diabetes.

The study evaluated and explored the effect of patient management and related factors under the Share Care management model aims to provide a clear evidence for the choice of new diagnosis and treatment strategies for patients with diabetes.

All patients enrolled in the study need to go through screening, initial visit, revisit, half-year visit and annual visit. The following is an overview of the research design.

Screening:

210 patients with type 2 diabetes who met the criteria were enrolled. All patients with informed consent will undergo basic interviews, vital sign measurements and related biochemical tests. During the screening phase, the following variables will be collected: age, sex, smoking status (current smokers, former smokers, non-smokers), duration of diabetes, duration of dyslipidemia, concomitant diseases and medication, etc. Besides, vital signs, 12-lead electrocardiogram, regular blood test and glycated hemoglobin (HbA1c), the patient's blood lipid spectrum includes total cholesterol (TC), triglyceride (TG), High density lipoprotein cholesterol (HDL-C) and low density lipoprotein cholesterol (LDL-C), albumin-to-creatinine ratio(ACR) and safety laboratory measurements (creatine kinase, SCr, BUN, UA, ALT, AST) also will be collected. The designated researcher will conduct a serum pregnancy test on all fertile women. The body mass index ((BMI)) is calculated by dividing weight by the square of height (kg / m2). After fasting overnight for 8 to 12 hours, the blood samples were collected before breakfast the next day. EGFR will be calculated using a Modification of diet in renal disease (MDRD).

Initial visit:

* Check the inclusion / exclusion criteria to confirm whether subjects are eligible to participate in the study. After confirming, the subjects will be randomly divided into the shared care group or the traditional therapy group according to the random number table.
* Basic vital signs: including height, weight, waist, hips, blood pressure, etc.
* Collection of metabolic indicators: HbA1c, ACR, blood biochemistry, etc.
* The number and days of emergency visits or hospitalizations due to diabetes-related factors (diabetic ketoacidosis, diabetic hyperosmotic coma, severe hypoglycemia) in the past three months before joining the study
* Filling in and recording the related behavior scale (summary of diabetes self-care activities (SDSCA), chinese diabetes management self-efficacy scale(C-DMSES), adjusted diabetes-specific quality of life scale (A-DQOL), morisky drug compliance scale and depression-anxiety-stress scale (DASS-21)).
* Insulin evaluation (including rotation of patients' insulin injection site, each change of needle, skin condition, preservation of insulin and correct use of insulin pen, etc.)
* Fundus evaluation.
* Foot evaluation.
* Health education.
* Daily medicine cost of patients

Revisit (every three months):

* Basic vital signs: including height, weight, waist, hips, blood pressure, etc.
* Collection of metabolic indicators: HbA1c, ACR, blood biochemistry, etc.
* The number and days of emergency visits or hospitalizations in the last three months (or since the last visit) due to diabetes-related factors (diabetic ketoacidosis, diabetic hyperosmotic coma, severe hypoglycemia)
* Daily medicine cost of patients half-year visit (every 6 months from the initial visit) needs to be added on the basis of the index of revisit.
* Basic vital signs: including height, weight, waist, hips, blood pressure, etc.
* Collection of metabolic indicators: HbA1c, ACR, blood biochemistry, etc.
* The number and days of emergency visits or hospitalizations in the last three months (or since the last visit) due to diabetes-related factors (diabetic ketoacidosis, diabetic hyperosmotic coma, severe hypoglycemia).
* Daily medicine cost of patients.
* Insulin evaluation.

Annual visit (every 12 months from the initial visit) in addition to all the indicators of revisit, there is also an increase:

* Filling in and recording the related behavior scale (summary of diabetes self-care activities (SDSCA), chinese diabetes management self-efficacy scale(C-DMSES), adjusted diabetes-specific quality of life scale (A-DQOL), morisky drug compliance scale and depression-anxiety-stress scale (DASS-21)).
* Insulin evaluation (including rotation of patients' insulin injection site, each change of needle, skin condition, preservation of insulin and correct use of insulin pen, etc.)
* Fundus evaluation.
* Foot evaluation.
* Insulin evaluation.

After being included in the study, patients were randomly divided into two groups: shared care group (experimental group) or traditional therapy group (control group). The total observation period for each patient was 1 year. Follow-up was carried out every 3 months. At each visit, the patient's basic condition, various vital signs and metabolic indicators, daily medicine cost of patients, and the number and days of emergency visits or hospitalizations in the last three months (or since the last visit) due to diabetes-related factors (diabetic ketoacidosis, diabetic hyperosmotic coma, severe hypoglycemia) will be collected.

Patients can download the Shared Care mobile application and connect with the smart-glucometer BG1 to upload blood glucose dairy in real time during the clinic. With patient's informed consent, the patient's follow-up data, laboratory indicators, etc. are uniformly collected and recorded for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years old diagnosed with type 2 diabetes
* Patients who have Informed and signed the consent form content
* Patients can be regularly followed (every 3 months) for at least 1 years

Exclusion Criteria:

* Patients with important organ failure or other severe diseases including infection, mentally disorder, heart failure or disseminated intravascular coagulation
* Patients with active or inactive malignant tumour, expectation of life less than 1 year
* Patients with communication disorders, cannot communicate and/or cooperate
* Females that are regnant, breast-feeding female, or conception plan in the recent year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic achieving rate | through study completion, 1 year follow-up
  Glycemic achieving rate with HbA1c<7% at 1-year follow-up

SECONDARY OUTCOMES:
HbA1c change | through study completion, 1 year follow-up
  Changes in HbA1c from baseline at 3, 6, and 12 months during follow-up
Blood pressure change and rate of reaching the standard | through study completion, 1 year follow-up
  Changes in blood pressure and the rate of reaching the standard (< 130/80) , including systolic blood pressure less than 130mmHg and diastolic blood pressure less than 80mmHg compared with the baseline at 3, 6, and 12 months respectively during follow-up.
LDL-c changes and rate of reaching the standard | through study completion, 1 year follow-up
  The changes of low density lipoprotein (LDL-c) compared with the baseline and the rate of reaching the standard (less than 2.6 mmol/L) at 3, 6, and 12 months during follow-up.
BMI change and rate of reaching the standard | through study completion, 1 year follow-up
  The changes of BMI from baseline and the rate of reaching the standard at 3, 6, and 12 months during follow-up. BMI is body mass index, weight and height will be combined to report BMI in kg/m^2
Medicine expenditure change | through study completion, 1 year follow-up
  Patients' daily medicine expenditure (rmb / day) changed from baseline at 3, 6, and 12 months during follow-up
SDSCA(Summary of Diabetes Self Care Activities) score change | through study completion, 1 year follow-up
  The change between baseline SDSCA score and SDSCA score 1 years after admission, SDSCA is scale Summary of Diabetes Self Care Activities (SDSCA), with 12 questions, each provide a minimum of 0 and maximum of 7 scores (7 indicates better self care action), total score 84.
C-DMSES(Chinese Diabetes Management Self-Efficacy Scale) score change | through study completion, 1 year follow-up
  The change between baseline C-DMSES and C-DMSES 1 years after admission. C-DMSES is Chinese Diabetes Management Self-Efficacy Scale. The scale measures the self-efficacy level of diabetes management. The C-DMSES has 20 questions, each question has a minimum score of 0 (indicates lowest self-efficacy), maximum score of 10(indicates highest self-efficacy). the scale has totally 200 scores.
A-DQOL(Amendment Diabetes Quality of Life scale) score change | through study completion, 1 year follow-up
  The change between baseline A-DQOL score and A-DQOL score 1 years after admission. CA-DQOL has maximum score of 230. Subscale 1 measures life satisfaction and has 15 questions, each question has a minimum score of 1 (indicates very unsatisfied), maximum score of 5(indicates very satisfied). Subscale 2 measures frequency of diabetes affects life quality, has 20 questions, each question has a minimum score of 1 (indicates never affect life quality), maximum score of 5(indicates always affect life quality). Subscale 3 measures how much the patient worries about how diabetes affects daily life and has 7 questions, each question has a minimum score of 1 (indicates never worries), maximum score of 5(indicates very worries). Subscale 4 measures how much the patient worries about the diabetes-related conditions and has 4 questions, each question has a minimum score of 1 (indicates never worries), maximum score of 5(indicates very worries).
Morisky scale score change | through study completion, 1 year follow-up
  The change between baseline Morisky score and Morisky score 1 years after admission. Morisky scale measures patients' compliance of medication usage. The Morisky scale has 4 questions, each question has a minimum score of 0 (did not comply the medical instruction), maximum score of 1(comply medical instruction). the scale has totally 4 scores.
DASS-C21 scale score change | through study completion, 1 year follow-up
  The change between baseline DASS-C21 scale score and DASS-C21 scale score 1 years after admission. DASS-C21 scale is Depression Anxiety Stress Scale 21 scale in Chinese. The scale measures patients' level of depression, anxiety and stress. The scale has 21 questions, each question has a minimum score of 0 (did not meet the description), maximum score of 3(completely meet the description). the scale has totally 63 scores.
Number of newly diagnosed diabetic complications | through study completion, 1 year follow-up
  During the follow-up period, number of newly diagnosed diabetic complications, including diabetic nephropathy, diabetic retinopathy, diabetic neuropathy and diabetic podiatry, etc.
The progress of diabetic complications | through study completion, 1 year follow-up
  During the follow-up period, the progress of diabetic complications such as diabetic nephropathy, diabetic retinopathy, diabetic neuropathy and diabetic foot disease
The times of Emergency visits due to hyperglycemia | through study completion, 1 year follow-up
  During the follow-up period, the times of Emergency visits due to hyperglycemia were collected during each follow-up.
The times of Emergency visits due to hypoglycemia | through study completion, 1 year follow-up
  During the follow-up period, the times of Emergency visits due to hypoglycemia were collected during each follow-up.
The times of Hospitalization due to hyperglycemia | through study completion, 1 year follow-up
  During the follow-up period, the times of hospitalization due to hyperglycemia were collected during each follow-up.
The times of Hospitalization due to hypoglycemia | through study completion, 1 year follow-up
  During the follow-up period, the times of hospitalization due to hypoglycemia were collected during each follow-up.
The days of Hospitalization due to hyperglycemia | through study completion, 1 year follow-up
  During the follow-up period, the days of hospitalization due to hyperglycemia were collected during each follow-up.
The days of Hospitalization due to hypoglycemia | through study completion, 1 year follow-up
  During the follow-up period, the days of hospitalization due to hypoglycemia were collected during each follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] International Diabetes Federation. IDF Diabetes Atlas. Brussels, Belgium: International Diabetes Federation 8th edition; 2017
- [Background] [A mass survey of diabetes mellitus in a population of 300,000 in 14 provinces and municipalities in China (author's transl)]. Zhonghua Nei Ke Za Zhi. 1981 Nov;20(11):678-83. No abstract available. Chinese. PMID 7341098
- [Background] Pan XR, Yang WY, Li GW, Liu J. Prevalence of diabetes and its risk factors in China, 1994. National Diabetes Prevention and Control Cooperative Group. Diabetes Care. 1997 Nov;20(11):1664-9. doi: 10.2337/diacare.20.11.1664. PMID 9353605
- [Background] Yang W, Lu J, Weng J, Jia W, Ji L, Xiao J, Shan Z, Liu J, Tian H, Ji Q, Zhu D, Ge J, Lin L, Chen L, Guo X, Zhao Z, Li Q, Zhou Z, Shan G, He J; China National Diabetes and Metabolic Disorders Study Group. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Mar 25;362(12):1090-101. doi: 10.1056/NEJMoa0908292. PMID 20335585
- [Background] Wang L, Gao P, Zhang M, Huang Z, Zhang D, Deng Q, Li Y, Zhao Z, Qin X, Jin D, Zhou M, Tang X, Hu Y, Wang L. Prevalence and Ethnic Pattern of Diabetes and Prediabetes in China in 2013. JAMA. 2017 Jun 27;317(24):2515-2523. doi: 10.1001/jama.2017.7596. PMID 28655017
- [Background] Ji LN, Lu JM, Guo XH, Yang WY, Weng JP, Jia WP, Zou DJ, Zhou ZG, Yu DM, Liu J, Shan ZY, Yang YZ, Hu RM, Zhu DL, Yang LY, Chen L, Zhao ZG, Li QF, Tian HM, Ji QH, Liu J, Ge JP, Shi LX, Xu YC. Glycemic control among patients in China with type 2 diabetes mellitus receiving oral drugs or injectables. BMC Public Health. 2013 Jun 21;13:602. doi: 10.1186/1471-2458-13-602. PMID 23800082
- [Background] Wan EYF, Fung CSC, Jiao FF, Yu EYT, Chin WY, Fong DYT, Wong CKH, Chan AKC, Chan KHY, Kwok RLP, Lam CLK. Five-Year Effectiveness of the Multidisciplinary Risk Assessment and Management Programme-Diabetes Mellitus (RAMP-DM) on Diabetes-Related Complications and Health Service Uses-A Population-Based and Propensity-Matched Cohort Study. Diabetes Care. 2018 Jan;41(1):49-59. doi: 10.2337/dc17-0426. Epub 2017 Nov 14. PMID 29138274
- [Background] American Diabetes Association. (11) Children and adolescents. Diabetes Care. 2015 Jan;38 Suppl:S70-6. doi: 10.2337/dc15-S014. No abstract available. PMID 25537712
- [Background] Type 2 diabetes in adults: management. London: National Institute for Health and Care Excellence (NICE); 2015 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK338142/ PMID 26741015
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness. JAMA. 2002 Oct 9;288(14):1775-9. doi: 10.1001/jama.288.14.1775. PMID 12365965
- [Background] Wagner EH, Grothaus LC, Sandhu N, Galvin MS, McGregor M, Artz K, Coleman EA. Chronic care clinics for diabetes in primary care: a system-wide randomized trial. Diabetes Care. 2001 Apr;24(4):695-700. doi: 10.2337/diacare.24.4.695. PMID 11315833
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555